CLINICAL TRIAL: NCT02682394
Title: Prognostic Importance of Quantitative Magnetic Resonance Imaging for Evaluation of Pancreatic Steatosis in Patients With Pancreatic Cancer
Brief Title: Evaluation of Pancreatic Steatosis in Patients With Cancer of Pancreas
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: SOR0216-15CTIL
Record Dates: First submitted 2015-12-28; First posted 2016-02-15 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2015-09

CONDITIONS: Cancer of Pancreas
Keywords: Cancer of pancreas; steatosis; MRI
MeSH Terms: conditions — Pancreatic Neoplasms; Fatty Liver

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cell-free DNA, CFD
Oversight: Data Monitoring Committee: No

SUMMARY:
Prognostic Importance of Quantitative Magnetic Resonance Imaging for Evaluation of Pancreatic Steatosis in Patients with Pancreatic Cancer

DETAILED DESCRIPTION:
1. Finding patients with pancreatic cancer (in all stages), before any treatment.
2. Non invasively quantify fatty infiltration of pancreas using, MRI DIXON Scan in pancreatic cancer patient relatively to liver.
3. Measuring cell-free blood DNA in those patients for evaluating the aggressiveness of the disease.
4. Quantify the prognostic significance of pancreatic steatosis in comparison with clinical and pathological prognostic indexes used today.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with any pancreatic cancer, in any stage, before treatment.
* >18 y.o

Exclusion Criteria:

* claustrophobia
* GFR<30
* patients with non mri compatible devices (e.g. orthopaedic external fixation system)
* After chemotherapy treatment or surgical procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 patients diagnosed with any pancreatic cancer, in any stage, before treatment.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-09 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of fat in pancreas measured in the head, body and tail excluding the lesion area. | at 24 hours before chemotherapy starting
  measuring Pancreatic Steatosis in patients with pancreatic cancer using MRI DIXON scan, at 24 hours before chemotherapy starting.
Blood levels of free DNA | The blood sample taken 15 minutes prior to MRI study, at time of IV access.
  Correlation of free DNA level and metastatic spread.

CONTACTS AND LOCATIONS:
Overall Officials: Alla Khashper, MD, Principal Investigator — Soroka University Medical Center
Locations (1):
- Soroka university medical center, Beersheba, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Ministry of Health, Israel. Israel Cancer Registry. — http://www.health.gov.il/UnitsOffice/HD/ICDC/ICR/CancerIncidence/Pages/default.aspx